CLINICAL TRIAL: NCT05840731
Title: Role of Ashwagandha Extract (Capsule KSM-66 300 mg) in Improving Sexual Health in Healthy Men: A Prospective, Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Role of Ashwagandha Extract (Capsule KSM-66 300 mg) in Improving Sexual Health in Healthy Men
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SF Research Institute, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Ixoreal-MSD-CT-01-22
Record Dates: First submitted 2023-04-14; First posted 2023-05-03 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: Sexual Health
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ashwagandha (Experimental): KSM-66 Ashwagandha is the active ingredient in Waithania somifera, a medicinal plant in Indian medicine. Ashwagandha is known as an adaptogen, an herb in capsule form that protects the body from stress.
  After enrollment in the study, 50% of participants will be randomly assigned to take one capsule of KSM 66 Ashwagandha (300 mg) two times daily after breakfast and every night at bedtime with food, preferably 30 minutes before the anticipated sexual intercourse with a glass of water for 8 weeks.
  Interventions: Dietary Supplement: Ashwagandha
- Placebo (Placebo Comparator): Placebo means that the capsules will not contain Ashwagandha but some other inactive substance. By using placebo, investigators will know whether the positive results are because of Ashwagandha or are because of psychological factors. For example, the participant may feel that his or her condition is improved because he or she is expecting the capsules to be helpful.
  After enrollment in the study, 50% of participants will be randomly assigned to take one capsule of placebo two times daily after breakfast and every night at bedtime with food, preferably 30 minutes before the anticipated sexual intercourse with a glass of water for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ashwagandha — KSM-66 Ashwagandha is the active ingredient in Waithania somifera, a medicinal plant in Indian medicine. Ashwagandha is known as an adaptogen, an herb in capsule form that protects the body from stress.
  Arms: Ashwagandha
Other: Placebo — Placebo means that the capsules will not contain Ashwagandha but some other inactive substance.
  Arms: Placebo

SUMMARY:
The clinical study aims to evaluate Efficacy and Safety of KSM66 Ashwagandha Standardized Root Extract for Improving Sexual Health in Healthy Men by measuring sex hormone levels in participant's blood, analyzing results of questionnaires, and monitoring adverse events in the post-marketing phase. Changes in the sex hormone levels in blood may affect sexual health or sexual health satisfaction. Efficacy is defined as increase in sex hormone levels in blood, and improvement in results or scores of assessment questionnaires.

DETAILED DESCRIPTION:
To qualify for this study, participant must be a healthy male between 30 to 50 years of age with unsatisfactory sexual health. Participants must NOT be taking medications or receiving treatments for erectile dysfunction. Participants are sexually active, and currently in a stable heterosexual relationship. Participants must agree to continue their routine diet and physical activities for the entire study. Participants should avoid using any NEW dietary supplements, multivitamins, or oral nutrition supplements throughout the study.

In this study, a maximum of 45 patients will be enrolled. The goal is to complete the study with at least 40 patients. At the initial visit, prospective patients will be screened for enrollment based on the requirements of the study, medical history, and clinical examination. Before starting any study related procedures, participants will be explained about the study in detail and a written informed consent will be obtained from participants prior to participation in this study. This document is a part of the written informed consent procedure. A detailed medical history including the associated conditions will be recorded. A general and physical examination will be performed to detect any abnormal parameters. If participants meet the eligibility criteria, they will be enrolled in the study.

After enrollment in the study, participants will be randomly assigned to take one capsule of KSM 66 Ashwagandha (300 mg) or one capsule of placebo two times daily after breakfast and every night at bedtime with food, preferably 30 minutes before the anticipated sexual intercourse with a glass of water for 8 weeks. There is a 50% chance that instead of 'Ashwagandha capsule' participants will receive 'Placebo capsule'. This placebo capsule will be identical in size, shape, and color to the 'Ashwagandha capsule'. The placebo capsule is harmless. It has the ingredient of starch powder made from corn, wheat, or potato. Participants will have to record the use of their assigned product on a daily diary for 8 weeks.

Participants will be monitored throughout the study. The study consists of two 60-minute onsite visits for visit 1 and visit 3, and one 40-minute remote visit via the phone for visit 2. After the initial visit 1 at the clinic (screening, baseline/randomization) (Day 1), participants will be monitored and assessed remotely at visit 2 (week 4) over the phone. Then, participants will have to come back to the clinic for assessments at visit 3 (week 8). During visit 1 and visit 3, blood will be collected from participants, physical examinations, and general examinations will be performed. During physical examinations, a medically trained personnel will measure participants' vital signs including systolic blood pressure, diastolic blood pressure, pulse rate, body temperature, respiratory rate, and body mass index. During general examination, a systemic review of different body systems will be performed to see if there are any significant abnormalities or findings.

For blood sample collection, participants' right or left arm will be used as the blood draw site. Investigators will take 12.5 ml of blood (less than the size of a tablespoon) from each participant to measure different sex hormone levels in his or her blood, such as dihydrotestosterone, follicle-stimulating hormone, luteinizing hormone, prolactin, and testosterone. Participants' blood samples will only be used for research and result analysis in this study. No more than 12.5 ml of blood will be drawn from each participant with a needle and syringe. All needles and syringes are brand new, and not recycled. All blood draws will be performed by professionally trained phlebotomists.

During remote visit 2 via phone, Satisfying Sexual Events (SSEs), Sexual Desire Inventory (SDI-2), International Index of Erectile Function (IIEF), Quality of Life (QoL) assessment questionnaires will be conducted over the phone. Side effects will be monitored, concomitant medications and study drug compliance will also be checked over the phone in visit 2.

At each visit, Satisfying Sexual Events (SSEs), Sexual Desire Inventory (SDI-2), International Index of Erectile Function (IIEF), Quality of Life (QoL) assessments will be conducted. Side effects will be monitored during each visit of the study period. Participants' results on all assessment questionnaires are confidential, and will only be reviewed by study staff, ethical review board members, and the FDA (if necessary). At visit 3 (week 8), participants are required to return any remaining testing products to the San Francisco Research Institute (at 2345 Ocean Ave, San Francisco, CA 94127) in person. Duration of the study is 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male participants between 30 to 50 years of age having poor sexual satisfaction based on his own perception since at least past 3 months.
* Participants whose IIEF-EF domain score is between 11 to 16 (i.e., moderately impaired).
* Participants in a stable, monogamous behavior and heterosexual relationship.
* Participants who are willing to stay away from any other medicines or treatments for Erectile Dysfunction (ED) during this study period.
* Participants who are willing to have 4 or more attempts of sexual intercourse each month.
* The participate should inform their partner about the study
* His partner should be willing to let him participate in the study
* Participants who are willing to take proper contraceptives during the study and within 3 months after the study completed. Proper contraceptives for participants include the following: (a) vasectomy (b) male condom with or without spermicide. Proper contraceptives for participant's partner include the following: (a) combined (estrogen and progesterone containing) hormonal contraception associated with inhibition of ovulation and/or implantation, such as oral birth control pills, intravaginal rings, or transdermal patches. (b) progesterone only hormonal contraception associated with inhibition of ovulation, such as oral pills, or injectable. (c) implantable progesterone only hormonal contraception associated with inhibition of ovulation and/or implantation, such as intrauterine device, intrauterine hormone releasing system. (d) bilateral tubal occlusion. (e) female condom with or without spermicide. (f) diaphragm with spermicide. (g) cervical cap with spermicide. (h) vaginal sponge with spermicide. (i) progesterone only oral hormonal contraception.
* Participants who have voluntarily decided to participate in this study and signed the informed consent form.
* Participants having sufficient understanding to communicate effectively with the investigator and are willing to discuss their sexual functioning with the investigative staff.
* Participants who are reliable, honest, compliant, and agree to co- operate with all trial evaluations as well as to be able to perform them as per investigator's opinion.
* Participants willing to follow the protocol requirements and agree to take an investigational product till 8 weeks ± 3 days.

Exclusion Criteria:

* Participants on any medication or supplement (e.g., ginseng, Sildenafil, vardenafil, tadalafil, avanafil) for improving the sexual function during the 3 months prior to study commencement.
* Participants having any clinically significant medical history, medical finding or an on-going medical or psychiatric condition or any acute illness which in the opinion of the Investigator could jeopardize the safety of the subject, impact validity of the study results or interfere with the completion of study according to the protocol.
* Individuals participating in any other studies, including macro/micro/any other forms of dietary supplements/multivitamins or disease-specific oral nutrition supplements (for improving the sexual function during the 3 months prior to study commencement).
* Participants having a history of hypersensitivity reactions (i.e., allergic or oversensitivity to usual doses).
* Participants with anatomical malformations of the penis.
* Participants with primary hypoactive sexual desire.
* Participants with ED, which is caused by any other primary sexual disorder, like hypopituitarism, hypothyroidism, or hypogonadism, hypergonadotropic.
* Participants who have a spinal injury or have had a radical prostatectomy.
* Participants with ED, which is caused by the failure of surgery in the pelvic cavity.
* Participants with penis deformity or penile implants.
* Participants with a history of malignancy.
* Participants with a major refractory psychiatric disorder or significant neurological abnormalities.
* Participants with alcohol addiction or persistent abuse of drugs of dependence.
* Partner of the participant is not planning to have pregnancy for next six months.
* Participants who are participating or discontinued participation in the past 3 months from any other clinical trial or are planning to father a baby or are in a relationship with a pregnant partner.

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2023-10-05 (Estimated); Study Completion 2023-10-12 (Estimated)

PRIMARY OUTCOMES:
Number of Satisfying Sexual Events (SSEs) | 8 weeks
  All enrolled subjects will be asked about SSEs 4 weeks prior Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1) and then throughout the study. It will include subject's inputs for number of intercourse and non-intercourse sexual events, number of orgasms, level of sexual desire, and satisfying sexual activity experienced.
  The subjects will be asked to mark a score for their sexual desire. They will be asked, "Indicate your most intense level of sexual desire in the last 24 hours/since your last visit." Potential responses included "no," "low," "moderate," or "strong", scored 0-3 (0 indicating no desire and 3 indicating the highest level of desire):
  0 = No desire
  1. = Low desire
  2. = Moderate desire
  3. = Strong desire
  Number of SSEs at Visit 3-End of study visit, (Week 8), will be compared with that of Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), and Visit 2 (Week 4).

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided